CLINICAL TRIAL: NCT06065007
Title: Quality of Life and Disease-related Symptoms in Individuals With Systemic Mastocytosis
Status: Active, not recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: SMQoL230918
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Mastocytosis, Systemic
MeSH Terms: conditions — Mastocytosis, Systemic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Swedish cohort of persons with Systemic Mastocytosis: We aim to include all individuals with a diagnosis of SM in Sweden, by identification via either one the two centers of excellence of mastocytosis or by a regional representative for the mastocytosis group in Sweden.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a cross-sectional observational study, no intervention will be implemented or exposure studied. Data for outcomes of interest will be collected via questionnaires

SUMMARY:
Systemic Mastocytosis is a rare and complex disease caused by accumulation of mast cells. The skin, bones, gastrointestinal tract, bone marrow and liver are the organs most often affected. Symptoms can vary greatly between patients. The study aims to describe the Swedish cohort's self-rated quality of life and levels of disease-related symptoms.

DETAILED DESCRIPTION:
Systemic Mastocytosis (SM) is a rare and complex disease caused by accumulation of mast cells leading to release of mediator substances (e.g., cytokines, prostaglandins, histamine and tryptase). The skin, bones, gastrointestinal tract, bone marrow and liver are the organs most often affected. Symptoms vary between patients and can include e.g., allergic reactions with anaphylaxis, rashes, osteoporoses, cognitive difficulties, fatigue, depression, anxiety, nausea, vomiting, stomach pains and diarrhea. In this cross-sectional observational study, the aim is to include the Swedish cohort of persons diagnosed with SM to gather a wide range of information on self-rated health-related quality of life, gastrointestinal symptoms, pain, anxiety, depression and self-care.

ELIGIBILITY:
Inclusion Criteria:

* Swedish-speaking individuals aged 18 years or older and diagnosed with indolent systemic mastocytosis (ISM) or advanced systemic mastocytosis (AdvSM), verified by a bone marrow biopsy

Exclusion Criteria:

* An assessment by the treating physician that the individual has a cognitive impairment making participation impossible
* The patient has undergone an allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with Systemic Masocytosis and meets the eligibility criteria, who are registered at one of the two existing mastocytosis centres in Sweden (Uppsala or Stockholm), or can be identified through a regional representative, will be asked to participate
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2028-11-15 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ C-30 | Day 1
  EORTC QLQ C-30 measures health related quality of life rated by individuals with malignancies and the general population. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems
The Mastocytosis Quality of Life Questionnaire (MC-QoL) | Day 1
  The Mastocytosis Quality of Life Questionnaire (MC-QoL), measures disease-specific quality of life items, has scores from 0 to 100, where higher scores indicate higher health-related quality-of-life impairment
The Hospital Anxiety and Depression Scale (HADS) | Day 1
  The Hospital Anxiety and Depression Scale (HADS), 14 items, is a screening tool for anxiety and depression in non-psychiatric clinical populations. There are 7 items for depression and 7 items for anxiety. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. A higher score indicates a higher level of distress.
The Gastrointestinal Symptom Rating Scale (GSRS) | Day 1
  The Gastrointestinal Symptom Rating Scale (GSRS), 15 items. This instrument measures The Gastrointestinal Symptom Rating Scale (GSRS). This instrument measures gastrointestinal symptoms in individuals with irritable bowel syndrome, gastric or duodenal ulcers and dyspepsia. The questionnaire, which contains 15 items, 6 subscales with total score between 19 to 133. Higher scores indicates more symptoms.
The Visceral Sensitivity Index (VSI) | Day 1
  The Visceral Sensitivity Index (VSI), 15 items, measures psychosocial consequences and worries of gastrointestinal symptoms. Each item scores 0-6 and a higher score indicates greater GI symptom-specific anxiety.
The Brief Pain Inventory - Short form (BPI-SF) | day 1
  The Brief Pain Inventory - Short form (BPI-SF), 9 items, yields a rating of levels of pain during a 24-hour period, and a description of the nature of that pain. The instrument also contains items on the impact (if any) of the pain of daily life. Each rating scale is bounded by the words "no pain" at the 0 end and "pain as bad as you can imagine" at the other. Using similar scales of 0 to 10, patients are also asked to rate the extent to which their pain interferes with 7 quality-of-life domains that include general activity, walking, mood, sleep, work, relations with other persons, and enjoyment of life. These scales are bounded by the words "does not interfere" and "interferes completely: Higher scores indicates higher levels of pain/Higher impact of pain on daily life.
The Brunnsviken Brief Quality of life scale (BBQ) | Day 1
  The Brunnsviken Brief Quality of life scale (BBQ), 12 items, has 4-graded response alternatives. The scale measures the overall self-experienced quality of life. The Satisfaction and Importance rating for each life area is multiplied and summed for a total quality of life score ((items 1 * 2) + (items 3 * 4) and so forth). Higher scores indicate higher levels of subjective QoL.
Self Care of Chronic Illness Inventory | Day 1
  Self Care of Chronic Illness Inventory, 29 items, measures self-care behaviors in persons with chronic illnesses. The scale measures three aspects of self care; Self-Care Maintenance, Self-Care Monitoring (or Symptom Perception), and Self-Care Management. Scores on each scale are standardized to range from 0 to100 with higher scores indicating better self-care

CONTACTS AND LOCATIONS:
Overall Officials: Mariann Hedström, PhD, Principal Investigator — Uppsala University, Department of Public Health and Caring Sciences
Locations (2):
- Sweden (2):
  - Karolinska Institutet, Stockholm
  - Uppsala University, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Anrooij B, Kluin-Nelemans JC, Safy M, Flokstra-de Blok BM, Oude Elberink JN. Patient-reported disease-specific quality-of-life and symptom severity in systemic mastocytosis. Allergy. 2016 Nov;71(11):1585-1593. doi: 10.1111/all.12920. Epub 2016 Jun 23. PMID 27089859
- [Background] Brockow K, Jofer C, Behrendt H, Ring J. Anaphylaxis in patients with mastocytosis: a study on history, clinical features and risk factors in 120 patients. Allergy. 2008 Feb;63(2):226-32. doi: 10.1111/j.1398-9995.2007.01569.x. PMID 18186813
- [Background] Fuchs D, Kilbertus A, Kofler K, von Bubnoff N, Shoumariyeh K, Zanotti R, Bonadonna P, Scaffidi L, Doubek M, Elberink HO, Span LFR, Hermine O, Elena C, Benvenuti P, Yavuz AS, Brockow K, Zink A, Aberer E, Gorska A, Romantowski J, Hadzijusufovic E, Fortina AB, Caroppo F, Perkins C, Illerhaus A, Panse J, Vucinic V, Jawhar M, Sabato V, Triggiani M, Parente R, Bergstrom A, Breynaert C, Gotlib J, Reiter A, Hartmann K, Niedoszytko M, Arock M, Kluin-Nelemans HC, Sperr WR, Greul R, Valent P. Scoring the Risk of Having Systemic Mastocytosis in Adult Patients with Mastocytosis in the Skin. J Allergy Clin Immunol Pract. 2021 Apr;9(4):1705-1712.e4. doi: 10.1016/j.jaip.2020.12.022. Epub 2020 Dec 23. PMID 33346151
- [Background] Gulen T, Hagglund H, Dahlen B, Nilsson G. Mastocytosis: the puzzling clinical spectrum and challenging diagnostic aspects of an enigmatic disease. J Intern Med. 2016 Mar;279(3):211-28. doi: 10.1111/joim.12410. Epub 2015 Sep 8. PMID 26347286
- [Background] Hermans MAW, Rietveld MJA, van Laar JAM, Dalm VASH, Verburg M, Pasmans SGMA, Gerth van Wijk R, van Hagen PM, van Daele PLA. Systemic mastocytosis: A cohort study on clinical characteristics of 136 patients in a large tertiary centre. Eur J Intern Med. 2016 May;30:25-30. doi: 10.1016/j.ejim.2016.01.005. Epub 2016 Jan 23. PMID 26809706
- [Background] Jennings S, Russell N, Jennings B, Slee V, Sterling L, Castells M, Valent P, Akin C. The Mastocytosis Society survey on mast cell disorders: patient experiences and perceptions. J Allergy Clin Immunol Pract. 2014 Jan-Feb;2(1):70-6. doi: 10.1016/j.jaip.2013.09.004. Epub 2013 Dec 3. PMID 24565772
- [Background] Jennings SV, Finnerty CC, Hobart JS, Martin-Martinez M, Sinclair KA, Slee VM, Agopian J, Akin C, Alvarez-Twose I, Bonadonna P, Bowman AS, Brockow K, Bumbea H, de Haro C, Fok JS, Hartmann K, Hegmann N, Hermine O, Kalisiak M, Katelaris CH, Kurz J, Marcis P, Mayne D, Mendoza D, Moussy A, Mudretzkyj G, Vaia NN, Niedoszytko M, Elberink HO, Orfao A, Radia DH, Rosenmeier S, Ribada E, Schinhofen W, Schwaab J, Siebenhaar F, Triggiani M, Tripodo G, Velazquez R, Wielink Y, Wimazal F, Yigit T, Zubrinich C, Valent P. Mast Cell Diseases in Practice and Research: Issues and Perspectives Raised by Patients and Their Recommendations to the Scientific Community and Beyond. J Allergy Clin Immunol Pract. 2022 Aug;10(8):2039-2051. doi: 10.1016/j.jaip.2022.06.018. Epub 2022 Jun 28. PMID 35777651
- [Background] Levedahl KH, Nilsson A, Ungerstedt J, Hedstrom M. Living with systemic mastocytosis: Balancing between vulnerability and resilience: A qualitative study. Eur J Oncol Nurs. 2022 Oct;60:102172. doi: 10.1016/j.ejon.2022.102172. Epub 2022 Jul 6. PMID 35963124
- [Background] Pardanani A. Systemic mastocytosis in adults: 2021 Update on diagnosis, risk stratification and management. Am J Hematol. 2021 Apr 1;96(4):508-525. doi: 10.1002/ajh.26118. Epub 2021 Feb 21. PMID 33524167
- [Background] Pulfer S, Ziehfreund S, Gebhard J, Hindelang B, Biedermann T, Brockow K, Zink A. Health-Related Quality of Life and Influencing Factors in Adults with Nonadvanced Mastocytosis-A Cross-Sectional Study and Qualitative Approach. J Allergy Clin Immunol Pract. 2021 Aug;9(8):3166-3175.e2. doi: 10.1016/j.jaip.2021.04.059. Epub 2021 May 26. PMID 33965596
- [Background] Siebenhaar F, von Tschirnhaus E, Hartmann K, Rabenhorst A, Staubach P, Peveling-Oberhag A, Wagner N, Martus P, Carter MC, Metcalfe DD, Church MK, Maurer M, Weller K. Development and validation of the mastocytosis quality of life questionnaire: MC-QoL. Allergy. 2016 Jun;71(6):869-77. doi: 10.1111/all.12842. Epub 2016 Feb 15. PMID 26797792
- [Background] Spolak-Bobryk N, Niedoszytko M, Jassem E, Chelminska M, Lange M, Majkowicz M, Nedoszytko B, Borchet J. The role of the clinical and psychological symptoms of mastocytosis in the patient's quality of life. Postepy Dermatol Alergol. 2022 Aug;39(4):688-696. doi: 10.5114/ada.2021.108433. Epub 2021 Sep 20. PMID 36090735
- [Background] Ungerstedt J, Ljung C, Klimkowska M, Gulen T. Clinical Outcomes of Adults with Systemic Mastocytosis: A 15-Year Multidisciplinary Experience. Cancers (Basel). 2022 Aug 16;14(16):3942. doi: 10.3390/cancers14163942. PMID 36010937
- [Derived] Hamberg Levedahl K, Carlson M, Nilsson GP, Jakobsson Larsson B, Ahsberg E, Hedstrom M. Investigating instruments for evaluation of gastrointestinal burdens in patients with systemic mastocytosis: an exploratory multimethod study. Scand J Gastroenterol. 2025 Dec 21:1-10. doi: 10.1080/00365521.2025.2604778. Online ahead of print. PMID 41424055